CLINICAL TRIAL: NCT03543020
Title: Radiation- Induced Alopecia in Patients Undergoing Radiation Therapy to the Brain: A Prospective Clinical and Dosimetric Study of Primary and Metastatic Brain Tumour Patients
Brief Title: Radiation- Induced Alopecia in Patients Undergoing Radiation Therapy to the Brain
Status: Terminated | Type: Observational
Why Stopped: inadequate patient number
Sponsor: Fortis Memorial Research Institute (Industry)
Responsible Party: Principal Investigator, Dr. Meena Mishra, Attending Consultant, Department of Radiation Oncology, Fortis Memorial Research Institute
Other Study IDs: 2017-008IP-20
Record Dates: First submitted 2018-05-16; First posted 2018-06-01 (Actual); Last update posted 2019-03-04 (Actual); Status verified 2019-03

CONDITIONS: Alopecia; X-Rays
Keywords: radiation induced alopecia; whole brain radiation; partial brain radiation; radiotherapy
MeSH Terms: conditions — Alopecia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients: Patients undergoing Radiation therapy to brain
  Interventions: Radiation: radiation therapy to brain

INTERVENTIONS:
Radiation: radiation therapy to brain — OSL placed over the scalp for initial 5 fractions for patients undergoing partial/ whole brain radiation therapy

SUMMARY:
Study will be conducted on patients receiving Whole brain(WB) / Partial Brain(PB) radiotherapy using volumetric modulated arc therapy or intensity modulated radiotherapy at Department of Radiation Oncology, Fortis Memorial Research Insititute, Gurgaon, Haryana with end points. 1) Primary - To observe degree of alopecia at conclusion of radiotherapy compared to pre- radiotherapy status using scalp sparing radiotherapy technique. 2) Secondary 1)Recording the temporal dose levels causing radiation associated alopecia and dose range acceptable for reversible radiation-induced alopecia and determine dose volume threshold for the same 2)Recording of scalp doses by in vivo dosimetry and correlation with radiation induced alopecia Methods: Study includes 50 patients of partial / whole brain radiation therapy to be followed consecutively for radiation- induced alopecia. Contouring: For WB radiation entire scalp will be contoured. For PB irradiation contouring of partial scalp to be done by drawing 2-3 cm beyond the PTV edge in all directions. Planning: The treatment planning and delivery to be done as per existing practice in department. Contouring at Monaco / Brain Lab Contouring stations and planning on Monaco Treatment planning system (TPS) Version 5.11.01. Duration: 18 months for patient accrual; in this observational study patients undergoing radiation therapy to brain will be evaluated clinically and objectively for degree of alopecia. Photographic and Clinical record of four views of scalp- Right lateral, Left lateral, top and rear to be taken at intervals- a)Pre-Radiotherapy (RT) b) RT Conclusion c) First follow-up at 1 month. Hair loss quantified using Severity of Alopecia Tool (SALT) Score. Dosimetric measurements having subcomponents - measurement of surface dose uses optically stimulated luminescence dosimeters to be placed over scalp for first 5 fractions in case of conventional or fractionated SRT, for the entire duration of short course treatments and for first 5 fractions in case of palliative whole brain radiation given over 10 fractions. TPS measurements: Average, maximum dose and dose per unit volume will be reported for whole and partial scalp. Outcomes 1. Quantify the degree of alopecia at the conclusion of radiotherapy as compared to pre- radiotherapy status. 2. To record the radiation dose levels causing alopecia. 3. Obtain in vivo dosimetry values for scalp doses in modern radiotherapy treatment

DETAILED DESCRIPTION:
Patients with primary or metastatic cancers to the brain need to undergo partial or whole brain radiotherapy. Alopecia is an inadvertent side effect of Radiation therapy to the brain. Much of this alopecia occurs in patches and is often associated with permanent loss of hair. Irradiation-induced epilation is due to high susceptibility of anagen follicles to radiation. Loss of hair can be stressful and distressing for cancer patients.

Various studies have tried to address the issue of threshold dose for radiotherapy induced alopecia. The severity and type of skin response and consequent alopecia to radiation is decided by multitude of factors - total dose and dose fractionation, quality of radiation, area or volume of tissue irradiated, anatomic site and vascular response. Studies have shown that 3Gy produces complete, reversible anagen alopecia and permanent alopecia begins to occur at 5Gy.

At higher dose rates the susceptibility of hair melanocytes is much more than epidermal melanocytes. Freysz et al in a retrospective analysis of 18 patients deduced that a cumulative dose as high as 12Gy results in alopecia that is reversible.Temporary alopecia is seen in most patients receiving WBRT with conventional fractionation. Most of these studies are either small reports or were done before the advent of modern technology. The advent of precision radiotherapy techniques has made it possible to utilize techniques that reduce the dose to the scalp in an attempt to minimize the chances of radiation- induced alopecia.

In a first, a phase II dosimetric and clinical study by De Puysseleyr et al concluded that Volumetric Modulated Arc Therapy (VMAT)- WBRT delivers lower scalp doses as compared to conventional parallel opposed fields but the study was closed prematurely as it failed to show any clinical benefit in terms of preventing alopecia. They however, concluded that the threshold Treatment Planning System (TPS) dose for temporary alopecia is around 10Gy in 5 fractions.

In a study by Ting et al alopecia was observed in half of the patients undergoing Whole Brain Radiotherapy (WBRT) to a dose of 30Gy/10 fractions did not have significant alopecia. The remaining half had mild alopecia. In the study by Mahadevan A et al, hippocampus sparing WBRT also spares hair follicle bearing regions of the scalp while maintaining strict compliance to hippocampus avoidance zone. There is no consensus regarding the threshold TPS dose for alopecia as the study of dose received by hair follicles during intensity modulated radiotherapy for whole brain is limited by lack of knowledge of dose-effect relation of temporary alopecia.

Rivero M et al have reported zero incidence of alopecia in the departmental protocol that they have developed for patients undergoing WBRT using 20Gy/5#s using SIB (40Gy/5#s) by VMAT. The different dose weightage and dose volumes practiced in their department have yielded excellent cosmetic outcomes.

The objective alopecia scoring scales have their own issues of inter-observer variability. EORTC BN20 questionnaire though a validated tool, is largely subjective. Since the expectation of a patient being treated by VMAT despite adequate counseling may be disproportionate to the reality of treatment outcomes, there may be marked deviation of scores to extremes. Severity of Alopecia Tool (SALT Score) is more objective with again the limitation of inter-observer variability. In order to minimize subjectivity, we will use SALT scoring system to analyze the degree of alopecia. SALT Score of 0 indicates no alopecia whereas score of 100 indicates complete baldness.

The investigators have been been using scalp contouring and scalp sparing radiotherapy technique to decrease the dose to the scalp with the aim to reduce alopecia.

This study aims to prospectively study the extent of alopecia by modern treatment techniques and assess the factors affecting the same.

Aims and Objectives:

This study will be conducted on patients receiving Whole brain radiotherapy (WBRT)/ Partial Brain RT using volumetric modulated arc therapy (VMAT) or intensity modulated radiotherapy (IMRT) at Radiation Oncology Department of FMRI, Gurgaon, Haryana with the following end points

Materials and Methods The study will include 50 patients undergoing partial / whole brain radiation therapy who will be assessed prospectively for radiation- induced alopecia.

Contouring: For whole brain radiation only, the whole scalp will be contoured. For partial brain irradiation contouring of lateral lesions partial scalp will be done. Partial scalp contouring shall be done by drawing 2-3 cm beyond the PTV edge in all directions. Partial scalp shall be considered as an organ at risk (OAR).

Planning: The treatment planning and treatment delivery of patients shall be done as per existing routine in the department. All contouring will be done at Monaco / BrainLab Contouring stations and planning will be done on Monaco Treatment planning system Version 5.11.01 using full or partial arc Volumetric modulated arc therapy (VMAT) technique. Patients treated by other techniques such as IMRT and 3-D CRT will also be included in this study and analysed. During radiotherapy planning dose constraints will be given without affecting the PTV coverage.

Following measurements shall be done -

1. Objective, Clinical and photographic analysis- Photographic and Clinical review record of the scalp(excluding the face of the patient) will include four views- Right lateral, Left lateral, top view and rear view of the scalp. These shall be done at following intervals- a) Before starting RT b) RT Conclusion c) First follow-up at 1 month. Hair loss will be quantified using the SALT Score. (14)
2. Dosimetric measurements: This shall have two subcomponents

   1. A measurement of surface dose uses optically stimulated luminescence (OSL) dosimeters that shall be placed over the scalp for first 5 fractions in case of conventional or fractionated Stereotactic Radiotherapy (SRT), for the entire duration of short course treatments and for first 5 fractions in case of palliative whole brain radiation given over 10 fractions. OSL will be placed on the scalp at the centre of arc span of the beams lateral and AP-PA views at the beam entry points. For reproducibility, OSL position will be marked on the Thermoplastic mask. Dose to OSL will be calculated after taking measurements during delivery of therapeutic dose.
   2. Treatment Planning system (TPS) measurements: In the TPS, the average, maximum dose and dose per unit volume will be reported for the whole scalp and partial scalp. In addition the routing measurements of dosimetry related to planning target volume(PTV) and organs at risk (OAR) shall be done as per existing norms

Statistical Methods Mean dose to the point of the OSL will be calculated from the Treatment planning system (TPS), and further the statistical co-relation between the measured and calculated dose will be evaluated by student t test using a 95% confidence interval. Mean scalp dose will be evaluated from the TPS. Further mean TPS calculated dose, measured dose and clinical outcome (degree of alopecia using SALT score) will be co-related using paired sample t test.

ELIGIBILITY:
Inclusion Criteria:

1. All patients with Central Nervous System tumors (primary/metastatic) undergoing radiation to whole brain/ partial brain.
2. All techniques of radiotherapy used for treatment delivery including VMAT and IMRT.
3. Fractionation regimes- conventional and hypofractionation.
4. Patients with KPS> 70, Patients able to communicate regarding the treatment side-effects.
5. Eligible patients willing to be a part of the trial.
6. Patients undergoing radiotherapy with or without concurrent Temozolomide

Exclusion Criteria:

1. Patients who have received prior radiotherapy to scalp.
2. Patients that need to be treated for scalp lesion such as squamous cell carcinomas of scalp.
3. Poor neurological status performance patients who are unable to communicate.
4. Prior co-morbidities/ dermatological conditions predisposing to pre-existent excessive hair fall (including Systemic Lupus Erythematosus, Hypothyroidism, Polycystic Ovarian Disease and similar conditions)
5. Patients unwilling to come for follow-up.
6. Patients who are completely bald.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients undergoing partial / whole brain radiation therapy in the Department of Radiation Oncology, Fortis Memorial Research Institute fulfiing the inclusion and exclusion criteria will be included in the study.
Sampling Method: Non-Probability Sample
Enrollment: 25 (Actual)
Dates: Start 2017-07-17 (Actual); Primary Completion 2018-12-31 (Actual); Study Completion 2019-01-30 (Actual)

PRIMARY OUTCOMES:
To record the degree of alopecia at the conclusion of radiotherapy compared to pre- radiotherapy status with use of scalp sparing radiotherapy technique. | From starting treatment to 1 month follow up post RT completion;
  To measure the alopecia at pre- RT, post RT completion and 1st follow up after 1 month of RT completion objectively using the SALT score.

SECONDARY OUTCOMES:
radiation dose range levels that causes alopecia | at 21 months
  to identify dose range levels that causes alopecia for every case
in vivo dosimetry values for scalp doses in modern radiotherapy treatment | first 5 days of radiation treatment
  to correlate the dose values of OSL with treatment planning system and assess the congruence between the two along with the dose range causing alopecia

CONTACTS AND LOCATIONS:
Overall Officials: Meena Mishra, M.D., Principal Investigator — Fortis Memorial Research Institute, Gurgaon, Haryana, India
Locations (1):
- Department of Radiation Oncology, Fortis Memorial Research Institute, Gurgaon, Haryana, India

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Auperin A, Arriagada R, Pignon JP, Le Pechoux C, Gregor A, Stephens RJ, Kristjansen PE, Johnson BE, Ueoka H, Wagner H, Aisner J. Prophylactic cranial irradiation for patients with small-cell lung cancer in complete remission. Prophylactic Cranial Irradiation Overview Collaborative Group. N Engl J Med. 1999 Aug 12;341(7):476-84. doi: 10.1056/NEJM199908123410703. PMID 10441603
- [Background] Slotman BJ, Mauer ME, Bottomley A, Faivre-Finn C, Kramer GW, Rankin EM, Snee M, Hatton M, Postmus PE, Collette L, Senan S. Prophylactic cranial irradiation in extensive disease small-cell lung cancer: short-term health-related quality of life and patient reported symptoms: results of an international Phase III randomized controlled trial by the EORTC Radiation Oncology and Lung Cancer Groups. J Clin Oncol. 2009 Jan 1;27(1):78-84. doi: 10.1200/JCO.2008.17.0746. Epub 2008 Dec 1. PMID 19047288
- [Background] Horton J, Baxter DH, Olson KB. The management of metastases to the brain by irradiation and corticosteroids. Am J Roentgenol Radium Ther Nucl Med. 1971 Feb;111(2):334-6. doi: 10.2214/ajr.111.2.334. No abstract available. PMID 5541678
- [Background] Batchelor D. Hair and cancer chemotherapy: consequences and nursing care--a literature study. Eur J Cancer Care (Engl). 2001 Sep;10(3):147-63. doi: 10.1046/j.1365-2354.2001.00272.x. PMID 11829374
- [Background] van Dijk IW, Cardous-Ubbink MC, van der Pal HJ, Heinen RC, van Leeuwen FE, Oldenburger F, van Os RM, Ronckers CM, Schouten-van Meeteren AY, Caron HN, Koning CC, Kremer LC. Dose-effect relationships for adverse events after cranial radiation therapy in long-term childhood cancer survivors. Int J Radiat Oncol Biol Phys. 2013 Mar 1;85(3):768-75. doi: 10.1016/j.ijrobp.2012.07.008. Epub 2012 Sep 3. PMID 22954771
- [Background] Steinmann D, Paelecke-Habermann Y, Geinitz H, Aschoff R, Bayerl A, Bolling T, Bosch E, Bruns F, Eichenseder-Seiss U, Gerstein J, Gharbi N, Hagg J, Hipp M, Kleff I, Muller A, Schafer C, Schleicher U, Sehlen S, Theodorou M, Wypior HJ, Zehentmayr F, van Oorschot B, Vordermark D. Prospective evaluation of quality of life effects in patients undergoing palliative radiotherapy for brain metastases. BMC Cancer. 2012 Jul 10;12:283. doi: 10.1186/1471-2407-12-283. PMID 22780988
- [Background] Bottomley A, Flechtner H, Efficace F, Vanvoorden V, Coens C, Therasse P, Velikova G, Blazeby J, Greimel E; European Organisation for Research and Treatment of Cancer (EORTC) Data Center and Quality of Life Group. Health related quality of life outcomes in cancer clinical trials. Eur J Cancer. 2005 Aug;41(12):1697-709. doi: 10.1016/j.ejca.2005.05.007. PMID 16043345
- [Background] Steinmann D, Schafer C, van Oorschot B, Wypior HJ, Bruns F, Bolling T, Sehlen S, Hagg J, Bayerl A, Geinitz H, Hipp M, Vordermark D. Effects of radiotherapy for brain metastases on quality of life (QoL). Prospective pilot study of the DEGRO QoL working party. Strahlenther Onkol. 2009 Mar;185(3):190-7. doi: 10.1007/s00066-009-1904-0. PMID 19330297
- [Background] De Puysseleyr A, Van De Velde J, Speleers B, Vercauteren T, Goedgebeur A, Van Hoof T, Boterberg T, De Neve W, De Wagter C, Ost P. Hair-sparing whole brain radiotherapy with volumetric arc therapy in patients treated for brain metastases: dosimetric and clinical results of a phase II trial. Radiat Oncol. 2014 Jul 29;9:170. doi: 10.1186/1748-717X-9-170. PMID 25074394
- [Background] Severs GA, Griffin T, Werner-Wasik M. Cicatricial alopecia secondary to radiation therapy: case report and review of the literature. Cutis. 2008 Feb;81(2):147-53. PMID 18441767
- [Background] Wen CS, Lin SM, Chen Y, Chen JC, Wang YH, Tseng SH. Radiation-induced temporary alopecia after embolization of cerebral arteriovenous malformations. Clin Neurol Neurosurg. 2003 Jul;105(3):215-7. doi: 10.1016/s0303-8467(03)00007-6. PMID 12860517
- [Background] Malkinson FD, Panizzon RG. Radiobiology and radiotherapy of skin diseases. In: Freedberg IM, Eisen AZ, Wolff K, Austen KF, Goldsmith LA, Katz SI, eds. Fitzpatricks dermatology in general medicine. 6th ed. New York: McGraw Hill Medical Publishing Division 2003; 1229-38.
- [Background] Freysz M, Mertz L, Lipsker D. [Temporary localized alopecia following neuroradiological procedures: 18 cases]. Ann Dermatol Venereol. 2014 Jan;141(1):15-22. doi: 10.1016/j.annder.2013.09.655. Epub 2013 Nov 7. French. PMID 24461089
- [Background] Gerrard GE, Prestwich RJ, Edwards A, Russon LJ, Richards F, Johnston CF, Kwok-Williams MC. Investigating the palliative efficacy of whole-brain radiotherapy for patients with multiple-brain metastases and poor prognostic features. Clin Oncol (R Coll Radiol). 2003 Oct;15(7):422-8. doi: 10.1016/s0936-6555(03)00148-1. PMID 14570092
- [Background] Mahadevan A, Sampson C, LaRosa S, Floyd SR, Wong ET, Uhlmann EJ, Sengupta S, Kasper EM. Dosimetric analysis of the alopecia preventing effect of hippocampus sparing whole brain radiation therapy. Radiat Oncol. 2015 Nov 26;10:245. doi: 10.1186/s13014-015-0555-9. PMID 26611656
- [Background] Mancini BR, Kim LH, Shaitelman SF, Yan D, Kestin LL, Grills IS: Intensity modulated or volumetric modulated radiation therapy (IMRT or VMAT) to reduce alopecia, xerostomia, and otitis after whole brain radiation therapy for brain metastases: a planning analysis. Int J Radiat Oncol Biol Phys 2010, 78: S840
- [Background] Roberge D, Parker W, Niazi TM, Olivares M. Treating the contents and not the container: dosimetric study of hair-sparing whole brain intensity modulated radiation therapy. Technol Cancer Res Treat. 2005 Oct;4(5):567-70. doi: 10.1177/153303460500400510. PMID 16173827
- [Background] Rivero M, Montero E, Ortiz M, Velazquez S, Dorado R. Avoidance of radiation induced alopecia en whole brain radiotherapy treatments with simultaneous integrated boost. Electronic Poster presentation at: 3rd ESTRO Forum; 2015 April 24-28; Barcelona, Spain; Elsevier; 2015, 115: S732-733
- [Background] Aaronson NK, Ahmedzai S, Bergman B, Bullinger M, Cull A, Duez NJ, Filiberti A, Flechtner H, Fleishman SB, de Haes JC, et al. The European Organization for Research and Treatment of Cancer QLQ-C30: a quality-of-life instrument for use in international clinical trials in oncology. J Natl Cancer Inst. 1993 Mar 3;85(5):365-76. doi: 10.1093/jnci/85.5.365. PMID 8433390
- [Background] Olsen EA, Hordinsky MK, Price VH, Roberts JL, Shapiro J, Canfield D, Duvic M, King LE Jr, McMichael AJ, Randall VA, Turner ML, Sperling L, Whiting DA, Norris D; National Alopecia Areata Foundation. Alopecia areata investigational assessment guidelines--Part II. National Alopecia Areata Foundation. J Am Acad Dermatol. 2004 Sep;51(3):440-7. doi: 10.1016/j.jaad.2003.09.032. No abstract available. PMID 15337988